CLINICAL TRIAL: NCT01309295
Title: A Prospective Study Evaluating the Efficacy and Safety of Mircera in Patients With CKD in Predialysis and Dialysis.
Brief Title: An Observational Study of Mircera (Methoxy Polyethylene Glycol-Epoetin Beta) in Patients With Chronic Kidney Disease in Pre-Dialysis or Dialysis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25465
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia, Kidney Disease, Chronic
MeSH Terms: conditions — Anemia; Kidney Diseases; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will assess the efficacy and safety of Mircera (methoxy polyethylene glycol-epoetin beta) in clinical practice in patients with chronic kidney disease, in pre-dialysis or on dialysis, initiated on Mircera treatment. Data from each patient will be collected over 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic kidney disease, in pre-dialysis or dialysis
* Appropriate for treatment with Mircera according to current guidelines and Summary of Product Characteristics

Exclusion Criteria:

* Anemia due to non-renal causes
* Pregnant or lactating women
* Uncontrolled hypertension
* Known hypersensitivity to methoxy polyethylene glycol-epoetin beta

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic kidney disease patients initiated on Mircera treatment
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Achievement of target hemoglobin (Hb) range of 10-12 g/dL according to Kidney Disease Outcomes Quality Initiative (KDQOI) guidelines | 2 years
Maintenance of target Hb range (10-12 g/dL) | 2 years
Safety: Incidence of adverse events | 2 years

SECONDARY OUTCOMES:
Correlation between baseline clinical variables and time on target Hb level | 2 years
Dosing pattern in clinical practice, including dose adaptations | 2 years
Frequency of visits and laboratory assessments | 2 years
Effect of compliance to treatment on Hb levels | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Tirana, Albania